CLINICAL TRIAL: NCT01922050
Title: Safety and Efficacy of Escalating Doses of Two LEO 43204 Formulations Applied Once Daily for Two Consecutive Days on Full Face or Approximately 250 cm2 (40 in2) on the Chest in Subjects With Actinic Keratosis
Brief Title: A Study of Increasing Strengths, Safety and Efficacy of Two Formulas of LEO 43204 on the Face or the Chest in Patients With Actinic Keratosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP0084-1013
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2019-02

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Part 1: LEO 43204 Formulation 1 (Experimental): Open-Label, Dose-Escalation, Once-Daily, 2-Day Treatment
  Interventions: Drug: LEO 43204 Formulation 1
- Part 1: LEO 43204 Formulation 2 (Experimental): Open-Label, Dose-Escalation, Once-Daily, 2-Day Treatment
  Interventions: Drug: LEO 43204 Formulation 2
- Part 2: LEO 43204 Formulation 1 Dose X (Experimental): Double-Blind, Once-Daily, 2-Day Treatment
  Interventions: Drug: LEO 43204 Formulation 1 Dose X
- Part 2: LEO 43204 Formulation 1 Dose Y (Experimental): Double-Blind, Once-Daily, 2-Day Treatment
  Interventions: Drug: LEO 43204 Formulation 1 Dose Y
- Part 2: LEO 43204 Formulation 2 Dose XX (Experimental): Double-Blind, Once-Daily, 2-Day Treatment
  Interventions: Drug: LEO 43204 Formulation 2 Dose XX
- Part 2: LEO 43204 Formulation 2 Dose YY (Experimental): Double-Blind, Once-Daily, 2-Day Treatment
  Interventions: Drug: LEO 43204 Formulation 2 Dose YY
- Part 2: Placebo Formulation 1 (Placebo Comparator): Double-Blind, Once-Daily, 2-Day Treatment
  Interventions: Drug: Placebo Formulation 1
- Part 2: Placebo Formulation 2 (Placebo Comparator): Double-Blind, Once-Daily, 2-Day Treatment
  Interventions: Drug: Placebo Formulation 2

INTERVENTIONS:
Drug: LEO 43204 Formulation 1
  Arms: Part 1: LEO 43204 Formulation 1
Drug: LEO 43204 Formulation 2
  Arms: Part 1: LEO 43204 Formulation 2
Drug: LEO 43204 Formulation 1 Dose X
  Arms: Part 2: LEO 43204 Formulation 1 Dose X
Drug: LEO 43204 Formulation 1 Dose Y
  Arms: Part 2: LEO 43204 Formulation 1 Dose Y
Drug: LEO 43204 Formulation 2 Dose XX
  Arms: Part 2: LEO 43204 Formulation 2 Dose XX
Drug: LEO 43204 Formulation 2 Dose YY
  Arms: Part 2: LEO 43204 Formulation 2 Dose YY
Drug: Placebo Formulation 1
  Arms: Part 2: Placebo Formulation 1
Drug: Placebo Formulation 2
  Arms: Part 2: Placebo Formulation 2

SUMMARY:
Part 1:

To identify Maximum Tolerated Dose (MTD) levels of two formulations of LEO 43204 after once daily treatment for two consecutive days

Part 2:

To evaluate efficacy of two formulations of LEO 43204 in two doses after once daily treatment for two consecutive days compared to vehicle formulations

ELIGIBILITY:
Inclusion Criteria:

1. Following verbal and written information about the trial, subject must provide informed consent documented by signing the Informed Consent Form (ICF) prior to any trial-related procedures.
2. Part 1: Subjects with 5 to 20 clinically typical, visible and discrete AKs on the face
3. Part 2: Subjects with 5 to 20 clinically typical, visible and discrete AKs on either the face or within a contiguous area of approximately 250 cm2 (40 in2) on the chest
4. Subject at least 18 years of age.
5. Female subjects must be of either:

   1. Non-childbearing potential, i.e., have a confirmed clinical history of sterility (e.g., the subject is without a uterus or have tubal ligation), or,
   2. Childbearing potential, provided there is a confirmed negative urine pregnancy test prior to trial treatment.
6. Female subjects of childbearing potential must use effective contraception throughout the study.

Exclusion Criteria:

1. Location of the treatment area within 5 cm (2 inches) of:

   1. an incompletely healed wound,
   2. a suspected basal or squamous cell carcinoma.
2. Prior treatment with ingenol mebutate gel on the treatment area.
3. Lesions in the treatment areas that have:

   1. atypical clinical appearance (e.g., hypertrophic, hyperkeratotic or cutaneous horns) and/or
   2. recalcitrant disease (e.g., did not respond to cryotherapy on two previous occasions).
4. History or evidence of skin conditions other than the trial indication that would interfere with the evaluation of the trial medication (e.g., eczema, unstable psoriasis, xeroderma pigmentosum, Rosacea), at the investigator's discretion.
5. Use of cosmetic or therapeutic products and procedures which could interfere with the assessments of the treatment areas.
6. Any other disease or medical condition such as history or presence of cancer, cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunological, or neurological disease or disorder, that, in the opinion of the investigator, makes the subject unsuitable to participate in the trial.
7. Any abnormal laboratory or ECG findings that are clinically significant and would impact the safety of the subjects or the interpretation of the study results, as determined by the investigator.
8. Anticipated need for hospitalisation or out-patient surgery during the first 15 days after the first trial medication application. Note that cosmetic/therapeutic procedures are not excluded if they fall outside of the criteria detailed in Prohibited Therapies or Medications.
9. Known sensitivity or allergy to any of the ingredients in the LEO 43204.
10. Presence of acute sunburn within the treatment areas.
11. Current enrolment or participation in an investigational clinical trial within 30 days of entry into this trial.
12. Subjects previously randomised in the trial (Part 1 or 2).
13. Female subjects who are breastfeeding.
14. In the opinion of the investigator, the subject is unlikely to comply with the Clinical Study Protocol (e.g., alcoholism, drug dependency or psychotic state).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Goldenberg, MD, Principal Investigator — Mount Sinai School of Medicine, Dermatology Faculty
Locations (25):
- United States (13):
  - Omni Dermatology, Phoenix, Arizona
  - Torrance Clinical Research Institute Inc., Lomita, California
  - Dermatology Cosmetic Laser Medical Associates of La Jolla, Inc., San Diego, California
  - Leavitt Medical Associates of Florida, Ormond Beach, Florida
  - Clinical Research Center, Morsani Center for Advanced Healthcare, Tampa, Florida
  - Research Institute of Deaconess Clinic, Evansville, Indiana
  - Hudson Dermatology, LLC, Evansville, Indiana
  - DermAssociates, PC, Rockville, Maryland
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Henry Ford Medical Center, Dept. of Dermatology, West Bloomfield, Michigan
  - The Dermatology Group, P.C., Verona, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Clinical Trials of Texas, Inc., San Antonio, Texas
- Canada (12):
  - Stratica Medical Inc., Edmonton, Alberta
  - Guildford Dermatology Specialists, Surrey, British Columbia
  - Durondel C.P. Inc./Dermatology Clinic, Moncton, New Brunswick
  - Ultranova Skincare, Barrie, Ontario
  - Co-Medica Research Network Inc., Courtice, Ontario
  - Dermatrials Research Incorporated, Hamilton, Ontario
  - The Guenther Dermatology Research Centre, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - XLR8 Medical Research, Windsor, Ontario
  - Centre de Recherche Dermatologique du Quebec Metropolitain, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bourcier M, Stein Gold L, Guenther L, Andreassen CM, Selmer J, Goldenberg G. A dose-finding trial with a novel ingenol derivative (ingenol disoxate: LEO 43204) for field treatment of actinic keratosis on full face or 250 cm2 on the chest. J Dermatolog Treat. 2017 Nov;28(7):652-658. doi: 10.1080/09546634.2017.1303568. Epub 2017 Apr 4. PMID 28264612

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: LEO 43204 Gel 0.0015: Part 1: Dose-Escalation
  LEO 43204 gel 0.0015% applied once daily for 2 consecutive days to full face or approximately 250 cm2 on the chest.
- Part 1: LEO 43204 Gel 0.003: Part 1: Dose-Escalation
  LEO 43204 gel 0.003% applied once daily for 2 consecutive days to full face or approximately 250 cm2 on the chest.
- Part 1: LEO 43204 Gel 0.006: Part 1: Dose-Escalation
  LEO 43204 gel 0.006% applied once daily for 2 consecutive days to full face or approximately 250 cm2 on the chest.
- Part 1: LEO 43204 Gel 0.012: Part 1: Dose-Escalation
  LEO 43204 gel 0.012% applied once daily for 2 consecutive days to full face or approximately 250 cm2 on the chest.
- Part 1: LEO 43204 Gel 0.018: Part 1: Dose-Escalation
  LEO 43204 gel 0.018% applied once daily for 2 consecutive days to full face or approximately 250 cm2 on the chest.
- Part 1: LEO 43204 Gel 0.025: Part 1: Dose-Escalation
  LEO 43204 gel 0.025% applied once daily for 2 consecutive days to full face or approximately 250 cm2 on the chest.
- Part 1: LEO 43204 Cream 0.0015: Part 1: Dose-Escalation
  LEO 43204 cream 0.0015% applied once daily for 2 consecutive days to full face or approximately 250 cm2 on the chest.
- Part 1: LEO 43204 Cream 0.003: Part 1: Dose-Escalation
  LEO 43204 cream 0.003% applied once daily for 2 consecutive days to full face or approximately 250 cm2 on the chest.
- Part 1: LEO 43204 Cream 0.006: Part 1: Dose-Escalation
  LEO 43204 cream 0.006% applied once daily for 2 consecutive days to full face or approximately 250 cm2 on the chest.
- Part 1: LEO 43204 Cream 0.012: Part 1: Dose-Escalation
  LEO 43204 cream 0.0012% applied once daily for 2 consecutive days to full face or approximately 250 cm2 on the chest.
- Part 2: LEO 43204 Gel 0.006: Part 2: Double-Blind phase
  LEO 43204 gel 0.006% applied once daily for 2 consecutive days to full face or approximately 250 cm2 on the chest. The first treatment was to be applied on Day 1 by the participant at the site under supervision of the study staff. The second treatment was applied by the participant on Day 2 at home.
- Part 2: LEO 43204 Gel 0.012: Part 2: Double-Blind phase LEO 43204 gel 0.012% applied once daily for 2 consecutive days to full face or approximately 250 cm2 on the chest. The first treatment was to be applied on Day 1 by the participant at the site under supervision of the study staff. The second treatment was applied by the participant on Day 2 at home.
- Part 2: LEO 43204 Gel 0.018: Part 2: Double-Blind phase LEO 43204 gel 0.018% applied once daily for 2 consecutive days to full face or approximately 250 cm2 on the chest. The first treatment was to be applied on Day 1 by the participant at the site under supervision of the study staff. The second treatment was applied by the participant on Day 2 at home.
- Part 2: LEO 43204 Gel Vehicle: Part 2: Double-Blind phase LEO 43204 gel vehicle applied once daily for 2 consecutive days to full face or approximately 250 cm2 on the chest. The first treatment was to be applied on Day 1 by the participant at the site under supervision of the study staff. The second treatment was applied by the participant on Day 2 at home.
Period: Part 1 Open-label, Dose-escalation Phase
Arm/Group | Part 1: LEO 43204 Gel 0.0015 | Part 1: LEO 43204 Gel 0.003 | Part 1: LEO 43204 Gel 0.006 | Part 1: LEO 43204 Gel 0.012 | Part 1: LEO 43204 Gel 0.018 | Part 1: LEO 43204 Gel 0.025 | Part 1: LEO 43204 Cream 0.0015 | Part 1: LEO 43204 Cream 0.003 | Part 1: LEO 43204 Cream 0.006 | Part 1: LEO 43204 Cream 0.012 | Part 2: LEO 43204 Gel 0.006 | Part 2: LEO 43204 Gel 0.012 | Part 2: LEO 43204 Gel 0.018 | Part 2: LEO 43204 Gel Vehicle
Started | 3 | 3 | 6 | 6 | 17 | 18 | 3 | 3 | 6 | 12 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 6 | 6 | 17 | 18 | 3 | 3 | 6 | 12 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 Double-blind Phase
Arm/Group | Part 1: LEO 43204 Gel 0.0015 | Part 1: LEO 43204 Gel 0.003 | Part 1: LEO 43204 Gel 0.006 | Part 1: LEO 43204 Gel 0.012 | Part 1: LEO 43204 Gel 0.018 | Part 1: LEO 43204 Gel 0.025 | Part 1: LEO 43204 Cream 0.0015 | Part 1: LEO 43204 Cream 0.003 | Part 1: LEO 43204 Cream 0.006 | Part 1: LEO 43204 Cream 0.012 | Part 2: LEO 43204 Gel 0.006 | Part 2: LEO 43204 Gel 0.012 | Part 2: LEO 43204 Gel 0.018 | Part 2: LEO 43204 Gel Vehicle
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 62 | 60 | 62 | 59
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 61 | 58 | 62 | 56
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are provided for all randomized participants
Groups:
- Part 1: LEO 43204 Gel 0.0015; Part 1: LEO 43204 Gel 0.003; Part 1: LEO 43204 Gel 0.006; Part 1: LEO 43204 Gel 0.012; Part 1: LEO 43204 Gel 0.018; Part 1: LEO 43204 Gel 0.025: Part 1: Open-Label, Dose-Escalation, Once-Daily, 2-Day Treatment
- Part 1: LEO 43204 Cream 0.0015; Part 1: LEO 43204 Cream 0.003; Part 1: LEO 43204 Cream 0.006; Part 1: LEO 43204 Cream 0.012: Part 1: Open-Label phase, Dose-Escalation, Once-Daily, 2-Day Treatment
- Part 2: LEO 43204 Gel Vehicle; Part 2: LEO 43204 Gel 0.006; Part 2: LEO 43204 Gel 0.012; Part 2: LEO 43204 Gel 0.018: Part 2: Double-Blind, Once-Daily, 2-Day Treatment
- Total: Total of all reporting groups
Arm/Group | Part 1: LEO 43204 Gel 0.0015 | Part 1: LEO 43204 Gel 0.003 | Part 1: LEO 43204 Gel 0.006 | Part 1: LEO 43204 Gel 0.012 | Part 1: LEO 43204 Gel 0.018 | Part 1: LEO 43204 Gel 0.025 | Part 1: LEO 43204 Cream 0.0015 | Part 1: LEO 43204 Cream 0.003 | Part 1: LEO 43204 Cream 0.006 | Part 1: LEO 43204 Cream 0.012 | Part 2: LEO 43204 Gel Vehicle | Part 2: LEO 43204 Gel 0.006 | Part 2: LEO 43204 Gel 0.012 | Part 2: LEO 43204 Gel 0.018 | Total
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 17 | 18 | 3 | 3 | 6 | 12 | 59 | 62 | 60 | 62 | 320
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 3 | 1 | 10 | 6 | 2 | 0 | 4 | 5 | 18 | 17 | 21 | 21 | 110
  >=65 years | 2 | 2 | 3 | 5 | 7 | 12 | 1 | 3 | 2 | 7 | 41 | 45 | 39 | 41 | 210
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 4 | 2 | 6 | 6 | 0 | 0 | 1 | 5 | 17 | 20 | 19 | 21 | 103
  Male | 2 | 2 | 2 | 4 | 11 | 12 | 3 | 3 | 5 | 7 | 42 | 42 | 41 | 41 | 217
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 32 | 31 | 31 | 32 | 126
  United States | 3 | 3 | 6 | 6 | 17 | 18 | 3 | 3 | 6 | 12 | 27 | 31 | 29 | 30 | 194

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants Experiencing a Dose Limiting Toxicity (DLT) Based on Local Skin Responses (LSRs)
Description: The number of participants experiencing DLTs are tabulated by treatment group. This was used to identify the maximum tolerated dose (MTD) of LEO 43204 after once daily treatment for 2 consecutive days.The MTD was defined as the highest dose level with less than 4 out of 12 participants(cohorts 1 to 4) or less than 6 out of 18 participants(cohorts 5 and 6) experiencing a DLT
  DLT was defined as one or more of the following 3 LSRs:
  * Crusting Grade 4
  * Erosion/Ulceration Grade 4
  * Vesiculation/Pustulation Grade 4
  or two or more of the following five LSRs:
  * Erythema Grade 4
  * Crusting Grade 3
  * Swelling Grade 4
  * Erosion/Ulceration Grade 3
  * Vesiculation/Pustulation Grade 3
  The Local Skin Responses consists of the following 6 categories: Erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, erosion/ulceration. Each individual LSR category are given a numeric grade of severity from 0-4. Grade 0 being no presence and 4 being the highest grade of severity.
Time Frame: From Day 1 up to and including Day 8
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Cohort 1: LEO 43204 Gel 0.0015; Part 1: Cohort 2: LEO 43204 Gel 0.003; Part 1: Cohort 3: LEO 43204 Gel 0.006; Part 1: Cohort 4: LEO 43204 Gel 0.012; Part 1: Cohort 5: LEO 43204 Gel 0.018; Part 1: Cohort 6: LEO 43204 Gel 0.025; Part 1: Cohort 1: LEO 43204 Cream 0.0015; Part 1: Cohort 2: LEO 43204 Cream 0.003; Part 1: Cohort 3: LEO 43204 Cream 0.006; Part 1: Cohort 4: LEO 43204 Cream 0.012: Part 1: Open-Label phase, Dose-Escalation, Once-Daily, 2-Day Treatment
Arm/Group | Part 1: Cohort 1: LEO 43204 Gel 0.0015 | Part 1: Cohort 2: LEO 43204 Gel 0.003 | Part 1: Cohort 3: LEO 43204 Gel 0.006 | Part 1: Cohort 4: LEO 43204 Gel 0.012 | Part 1: Cohort 5: LEO 43204 Gel 0.018 | Part 1: Cohort 6: LEO 43204 Gel 0.025 | Part 1: Cohort 1: LEO 43204 Cream 0.0015 | Part 1: Cohort 2: LEO 43204 Cream 0.003 | Part 1: Cohort 3: LEO 43204 Cream 0.006 | Part 1: Cohort 4: LEO 43204 Cream 0.012
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 17 | 18 | 3 | 3 | 6 | 12
Participants
  No | 3 | 3 | 6 | 6 | 17 | 12 | 3 | 3 | 6 | 9
  Yes | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 3

2. Primary Outcome: Part 2: Percent Reduction From Baseline in Actinic Keratosis (AK) Counts (Multiple Imputation)
Time Frame: At Week 8
Population: The analysis was based on the Full Analysis Set, which was defined as all randomized participants who applied investigation product. One participant from the LEO 43204 gel vehicle arm did not apply investigation product, and thus was excluded from the efficacy analysis.
Measure: Mean (95% Confidence Interval); unit: percentage of reduction
Arm/Group | Part 2: LEO 43204 Gel Vehicle | Part 2: LEO 43204 Gel 0.006 | Part 2: LEO 43204 Gel 0.012 | Part 2: LEO 43204 Gel 0.018
Number analyzed (Participants) | 58 | 62 | 60 | 62
percentage of reduction | 42.3 [30.5 to 52.1] | 69.7 [63.1 to 75.1] | 73.4 [67.1 to 78.5] | 79.0 [74.0 to 83.0]
Statistical Analysis 1: Comparison: Part 2: LEO 43204 Gel Vehicle vs Part 2: LEO 43204 Gel 0.006; Test type: Superiority; p < 0.001, Negative binominal regression; Negative binominal regression with log baseline count as offset variable and treatment group and analysis site as factors; Rate ratio = 0.53, 95% CI 2-sided [0.40 to 0.69]
Statistical Analysis 2: Comparison: Part 2: LEO 43204 Gel Vehicle vs Part 2: LEO 43204 Gel 0.012; Test type: Superiority; p < 0.001, Negative binominal regression; [statistical method as in outcome 2, analysis 1]; Rate ratio = 0.46, 95% CI 2-sided [0.35 to 0.61]
Statistical Analysis 3: Comparison: Part 2: LEO 43204 Gel Vehicle vs Part 2: LEO 43204 Gel 0.018; Test type: Superiority; p < 0.001, Negative binominal regression; [statistical method as in outcome 2, analysis 1]; Rate ratio = 0.36, 95% CI 2-sided [0.28 to 0.48]
Statistical Analysis 4: Comparison: Part 2: LEO 43204 Gel 0.006 vs Part 2: LEO 43204 Gel 0.012; Test type: Superiority; p = 0.38, Negative binominal regression; [statistical method as in outcome 2, analysis 1]; Rate ratio = 0.88, 95% CI 2-sided [0.66 to 1.17]
Statistical Analysis 5: Comparison: Part 2: LEO 43204 Gel 0.006 vs Part 2: LEO 43204 Gel 0.018; Test type: Superiority; p = 0.013, Negative binominal regression; [statistical method as in outcome 2, analysis 1]; Rate ratio = 0.69, 95% CI 2-sided [0.52 to 0.93]
Statistical Analysis 6: Comparison: Part 2: LEO 43204 Gel 0.012 vs Part 2: LEO 43204 Gel 0.018; Test type: Superiority; p = 0.13, Negative binominal regression; [statistical method as in outcome 2, analysis 1]; Rate ratio = 0.79, 95% CI 2-sided [0.58 to 1.07]

3. Secondary Outcome: Part 2: Percentage of Participants With Complete Clearance of Actinic Keratosis Lesions (AKs) (Multiple Imputation)
Description: Complete clearance was defined as a 100% reduction from baseline in AK count. For treatment groups Vehicle, 0.006 and 0.012 the table shows the percentage of mean number of participants across imputations with complete clearance. For treatment group 0.018 the table shows the percentage of mean number of participants with complete clearance in observed cases.
Time Frame: At Week 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: LEO 43204 Gel Vehicle | Part 2: LEO 43204 Gel 0.006 | Part 2: LEO 43204 Gel 0.012 | Part 2: LEO 43204 Gel 0.018
Number analyzed (Participants) | 58 | 62 | 60 | 62
percentage of participants | 12.2 [3.7 to 20.7] | 9.9 [2.4 to 17.3] | 18.8 [8.8 to 28.8] | 24.2 [13.5 to 34.9]
Statistical Analysis 1: Comparison: Part 2: LEO 43204 Gel Vehicle vs Part 2: LEO 43204 Gel 0.006; Log binomial regression with treatment group as factor and baseline AK count included as covariate; Test type: Superiority; p = 0.57, Log binomial regression; Ratio of clearance rates = 0.74, 95% CI 2-sided [0.27 to 2.04]
Statistical Analysis 2: Comparison: Part 2: LEO 43204 Gel Vehicle vs Part 2: LEO 43204 Gel 0.012; Log binomial regression with treatment group as factor and baseline AK count included as covariate; Test type: Superiority; p = 0.51, Log binomial regression; Ratio of clearance rates = 1.33, 95% CI 2-sided [0.56 to 3.13]
Statistical Analysis 3: Comparison: Part 2: LEO 43204 Gel Vehicle vs Part 2: LEO 43204 Gel 0.018; Log binomial regression with treatment group as factor and baseline AK count included as covariate; Test type: Superiority; p = 0.11, Log binomial regression; Ratio of clearance rates = 1.90, 95% CI 2-sided [0.86 to 4.21]
Statistical Analysis 4: Comparison: Part 2: LEO 43204 Gel 0.006 vs Part 2: LEO 43204 Gel 0.012; Log binomial regression with treatment group as factor and baseline AK count included as covariate; Test type: Superiority; p = 0.21, Log binomial regression; Ratio of clearance rates = 1.79, 95% CI 2-sided [0.72 to 4.43]
Statistical Analysis 5: Comparison: Part 2: LEO 43204 Gel 0.006 vs Part 2: LEO 43204 Gel 0.018; Log binomial regression with treatment group as factor and baseline AK count included as covariate; Test type: Superiority; p = 0.031, Log binomial regression; Ratio of clearance rates = 2.55, 95% CI 2-sided [1.09 to 5.98]
Statistical Analysis 6: Comparison: Part 2: LEO 43204 Gel 0.012 vs Part 2: LEO 43204 Gel 0.018; Log binomial regression with treatment group as factor and baseline AK count included as covariate; Test type: Superiority; p = 0.29, Log binomial regression; Ratio of clearance rates = 1.43, 95% CI 2-sided [0.74 to 2.75]

4. Secondary Outcome: Part 2: Percentage of Participants With Partial Clearance of AKs (Multiple Imputation)
Description: Partial clearance was defined as at least 75% reduction from baseline in AK count.
  For treatment groups Vehicle, 0.006 and 0.012 the table shows the percentage of mean number of participants across imputations with partial clearance. For treatment group 0.018 the table shows the percentage of mean number of participants with partial clearance in observed cases.
Time Frame: At Week 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: LEO 43204 Gel Vehicle | Part 2: LEO 43204 Gel 0.006 | Part 2: LEO 43204 Gel 0.012 | Part 2: LEO 43204 Gel 0.018
Number analyzed (Participants) | 58 | 62 | 60 | 62
percentage of participants | 29.9 [18.0 to 41.9] | 52.4 [39.9 to 64.9] | 54.5 [41.8 to 67.2] | 62.9 [50.9 to 74.9]
Statistical Analysis 1: Comparison: Part 2: LEO 43204 Gel Vehicle vs Part 2: LEO 43204 Gel 0.006; Log binomial regression with treatment group as factor and baseline AK count included as covariate; Test type: Superiority; p = 0.026, Log binomial regression; Ratio of clearance rates = 1.69, 95% CI 2-sided [1.06 to 2.69]
Statistical Analysis 2: Comparison: Part 2: LEO 43204 Gel Vehicle vs Part 2: LEO 43204 Gel 0.012; Log binomial regression with treatment group as factor and baseline AK count included as covariate; Test type: Superiority; p = 0.013, Log binomial regression; Ratio of clearance rates = 1.79, 95% CI 2-sided [1.13 to 2.84]
Statistical Analysis 3: Comparison: Part 2: LEO 43204 Gel Vehicle vs Part 2: LEO 43204 Gel 0.018; Test type: Superiority; p < 0.001, Log binomial regression; Ratio of clearance rates = 2.10, 95% CI 2-sided [1.35 to 3.25]
Statistical Analysis 4: Comparison: Part 2: LEO 43204 Gel 0.006 vs Part 2: LEO 43204 Gel 0.012; Test type: Superiority; p = 0.73, Log binomial regression; Ratio of clearance rates = 1.06, 95% CI 2-sided [0.76 to 1.47]
Statistical Analysis 5: Comparison: Part 2: LEO 43204 Gel 0.006 vs Part 2: LEO 43204 Gel 0.018; Test type: Superiority; p = 0.16, Log binomial regression; Ratio of clearance rates = 1.24, 95% CI 2-sided [0.92 to 1.67]
Statistical Analysis 6: Comparison: Part 2: LEO 43204 Gel 0.012 vs Part 2: LEO 43204 Gel 0.018; Log binomial regression with treatment group as factor and baseline AK count included as covariate; Test type: Superiority; p = 0.30, Log binomial regression; Ratio of clearance rates = 1.17, 95% CI 2-sided [0.87 to 1.57]

ADVERSE EVENTS:
Time Frame: From Day 1 to Week 8
Description: The safety analysis was based on the Safety Analysis Set, which was defined as all randomized participants who received at least 1 application of investigational product and had safety information available post treatment. One participant from the LEO 43204 gel vehicle arm did not apply investigation product, and this was excluded from the safety analysis.
Arm/Group | Part 1: LEO 43204 Gel 0.0015 | Part 1: LEO 43204 Gel 0.003 | Part 1: LEO 43204 Gel 0.006 | Part 1: LEO 43204 Gel 0.012 | Part 1: LEO 43204 Gel 0.018 | Part 1: LEO 43204 Gel 0.025 | Part 1: LEO 43204 Cream 0.0015 | Part 1: LEO 43204 Cream 0.003 | Part 1: LEO 43204 Cream 0.006 | Part 1: LEO 43204 Cream 0.012 | Part 2: LEO 43204 Gel Vehicle | Part 2: LEO 43204 Gel 0.006 | Part 2: LEO 43204 Gel 0.012 | Part 2: LEO 43204 Gel 0.018
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/6 | 0/6 | 1/17 | 0/18 | 0/3 | 0/3 | 0/6 | 0/12 | 0/58 | 5/62 | 2/60 | 0/62
Other Adverse Events (participants affected / at risk) | 3/3 | 1/3 | 5/6 | 5/6 | 10/17 | 11/18 | 1/3 | 1/3 | 2/6 | 8/12 | 11/58 | 38/62 | 40/60 | 47/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: LEO 43204 Gel 0.0015 (N=3) | Part 1: LEO 43204 Gel 0.003 (N=3) | Part 1: LEO 43204 Gel 0.006 (N=6) | Part 1: LEO 43204 Gel 0.012 (N=6) | Part 1: LEO 43204 Gel 0.018 (N=17) | Part 1: LEO 43204 Gel 0.025 (N=18) | Part 1: LEO 43204 Cream 0.0015 (N=3) | Part 1: LEO 43204 Cream 0.003 (N=3) | Part 1: LEO 43204 Cream 0.006 (N=6) | Part 1: LEO 43204 Cream 0.012 (N=12) | Part 2: LEO 43204 Gel Vehicle (N=58) | Part 2: LEO 43204 Gel 0.006 (N=62) | Part 2: LEO 43204 Gel 0.012 (N=60) | Part 2: LEO 43204 Gel 0.018 (N=62)
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: LEO 43204 Gel 0.0015 (N=3) | Part 1: LEO 43204 Gel 0.003 (N=3) | Part 1: LEO 43204 Gel 0.006 (N=6) | Part 1: LEO 43204 Gel 0.012 (N=6) | Part 1: LEO 43204 Gel 0.018 (N=17) | Part 1: LEO 43204 Gel 0.025 (N=18) | Part 1: LEO 43204 Cream 0.0015 (N=3) | Part 1: LEO 43204 Cream 0.003 (N=3) | Part 1: LEO 43204 Cream 0.006 (N=6) | Part 1: LEO 43204 Cream 0.012 (N=12) | Part 2: LEO 43204 Gel Vehicle (N=58) | Part 2: LEO 43204 Gel 0.006 (N=62) | Part 2: LEO 43204 Gel 0.012 (N=60) | Part 2: LEO 43204 Gel 0.018 (N=62)
Application site pain (General disorders) | 1 | 1 | 2 | 3 | 3 | 8 | 0 | 1 | 0 | 5 | 5 | 25 | 33 | 37
Application site pruritus (General disorders) | 1 | 1 | 2 | 4 | 2 | 1 | 0 | 0 | 0 | 4 | 1 | 14 | 14 | 16
Application site erythema (General disorders) | 0 | 0 | 2 | 1 | 2 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Application site discolouration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 2 | 6
Application site exfoliation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Application site photosensitivity reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2
Scintillating scotoma (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 6 | 5
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Application site warmth (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site paraesthesia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2
Application site dermatitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Application site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Application site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Granuloma skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigator's right to publish the entire results of the study, irrespective of outcome. LEO retains the right to have any publication submitted to LEO for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.